CLINICAL TRIAL: NCT04419155
Title: ESCAP-2020-CPHG: Treatment Strategies Follow-up Implemented During the First Three Years Following Primary Lung Cancer (PLC) Diagnosed in KBP-2020-CPHG Cohort Patients
Acronym: ESCAP-2020
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Collège des Pneumologues des Hôpitaux Généraux (Other)
Responsible Party: Sponsor
Other Study IDs: A00943-54
Record Dates: First submitted 2020-04-27; First posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prognosis for primary lung cancer (PLC) is very limited. In France, patients diagnosed for PLC in 2010 and followed in Respiratory Medicine or Oncology department of a General Hospital Centre had a 5-year survival rate of 12.7% (vs 10% in 2000).

Over the last ten years, substantial improvements have been made both in terms of diagnostic (immunohistochemistry and molecular biology) and therapeutic. New treatments have been marketed and are now available in clinic.

New therapeutical strategies have been launched and have proved their efficacy in clinical studies or meta-analyses, generally increasing the survival rate of patients by a few months. However, little information still exists on the use and effectiveness of these molecules in clinical practice.

The CPHG proposes to complete the information collected during KPB-2020-CPHG study by the ESCAP-2020-CPHG study that is a follow-up of therapeutical strategies over the first 3 years of treatment. This study should improve knowledge of the PLC treatment management in General Hospital Centres.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Primary Lung Cancer histologically (or cytologically or presence of a mutation on liquid biopsy with compatible imaging) proven between January 1st and December 31st, 2020*
* Follow-up by a lung specialist at a General Hospital
* Oral informed consent * date of collected sample

Exclusion Criteria:

* Age < 18 years
* Secondary lung cancer
* Recurrence of same histological type PLC- left to the investigator discretion according to the clinic and the imagery
* Previous enrolment in the study
* Freedom deprived patient following a legal or administrative decision
* Patient unable to give his(her) consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Primary Lung Cancer histologically or cytologically proven between January 1st and December 31st, 2020
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Describe therapeutical strategies implemented by pulmonologists in Respiratory Medicine or Oncology department of a General Hospital Centres during the first three years following PLC diagnosed in KBP-2020-CPHG cohort patients. | 3 years
  Data collected for the ESCAP-2020-CPHG study:
  - All treatments administered

CONTACTS AND LOCATIONS:
Locations (1):
- Collège des Pneumologues des Hôpitaux Généraux (CPHG) (General Hospital Pulmonologists College), Paris, France

IPD SHARING:
Plan to Share IPD: No